CLINICAL TRIAL: NCT03705221
Title: Healthy Parent Carers Programme: Feasibility Study of a Peer-led Group-based Health Promotion Intervention for Parent Carers of Disabled Children Using a Parallel Group Randomised Controlled Trial Design
Brief Title: Healthy Parent Carers Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NIHR RfPB PB-PG-0317-20044; 246169 (Other: IRAS)
Record Dates: First submitted 2018-10-10; First posted 2018-10-15 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group programme (Experimental): Healthy Parent Carers group programme: A group-based peer led manualised programme called Healthy Parent Carers. The programme content is organised into 12 modules, which can be delivered over six longer (4-hour) sessions or 12 shorter (2-hour) sessions.
  Interventions: Behavioral: Healthy Parent Carers group programme
- Online resources (Active Comparator): Healthy Parent Carers online resources: Online resources from the Healthy Parent Carers programme, including materials for 12 modules and related videos and audio files to illustrate the content.
  Interventions: Behavioral: Healthy Parent Carers online resources

INTERVENTIONS:
Behavioral: Healthy Parent Carers group programme — Peer-led group-based weekly programme.
  Arms: Group programme
Behavioral: Healthy Parent Carers online resources — Online resources related to health and wellbeing
  Arms: Online resources

SUMMARY:
This study is a feasibility study of a peer-led group-based health promotion intervention for parent carers. It will used a parallel group randomised controlled trial design to compare a group based intervention called Healthy Parent Carers, with online resources about improving health and wellbeing.

DETAILED DESCRIPTION:
The objectives of the study are:

1. to evaluate whether the programme can be delivered in the community, and
2. to provide information necessary to design a definitive randomised controlled trial.

The investigators aim to recruit at least 96 parent carers of children with special educational needs and disabilities aged up to 25 years in six sites in Devon, Cornwall and Somerset. Participants will be individually randomised, stratified by group delivery site when recruitment in each site is completed, to either take part in a group programme, which includes online Healthy Parent Carer programme materials (intervention), or to receive access to the online materials for self-study only (control).

The programme content is organised into 12 modules, which can be delivered over six longer (4-hour) sessions or 12 shorter (2-hour) sessions. Groups will consist of at least 6 parent carers. The participant materials will be provided online.

Demographics will be collected at baseline. Participants will complete measures of mental health, wellbeing, health-related quality of life, health behaviours, patient activation, protective factors, and resource use. These data will be collected before randomisation (baseline), at post-intervention (i.e. after the intervention arm completes the group programme), and at 6 months post-intervention.

Recruitment will be monitored in order to plan for a definitive trial. Facilitators' adherence to the Facilitator Manual and participant engagement will be monitored using a facilitator checklist at the end of the sessions and we will audio-record the training sessions and group sessions. Participants' will provide feedback on the programme to assess the acceptability of the outcome measures. The investigators will conduct interviews with a sample of participants in both study arms and a focus group with facilitators to provide insights into intervention content, delivery and experience.

ELIGIBILITY:
Inclusion Criteria:

* a) Primary carers of children who identify that their children have additional needs and/or disabilities. Participants who self-identify as primary carers are eligible. The child should be up to 25 years old (this age range is consistent with the current UK Department of Health and Department of Education Special Educational Needs & Disability (SEND) legislation and The Children's Act);

  b) Willing and able to attend the programme group meeting session(s) on arranged dates/times;

  c) Able to access online information.

Exclusion Criteria:

* a) Not able to communicate in English.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-02-04 (Actual); Study Completion 2020-02-04 (Actual)

PRIMARY OUTCOMES:
Warwick-Edinburgh Mental Well-being Scale | 6 months post-intervention
  The Warwick-Edinburgh Mental Well-being Scale (WEMWBS) is a 14-item scale used to assess mental wellbeing in the general population and in evaluation of programmes aiming to improve mental wellbeing.

SECONDARY OUTCOMES:
Warwick-Edinburgh Mental Well-being Scale | Baseline
  The Warwick-Edinburgh Mental Well-being Scale (WEMWBS) is a 14-item scale used to assess mental wellbeing in the general population and in evaluation of programmes aiming to improve mental wellbeing.
Warwick-Edinburgh Mental Well-being Scale | Immediately post-intervention (up to 12 weeks)
  The Warwick-Edinburgh Mental Well-being Scale (WEMWBS) is a 14-item scale used to assess mental wellbeing in the general population and in evaluation of programmes aiming to improve mental wellbeing.
EQ-5D-5L | Baseline
  The EuroQol-5 Dimensions (EQ-5D-5L) is a measure of health-related quality of life. It consists of five items measuring five dimensions of health-related quality of life (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a vertical visual analogue scale measuring self-rated health.
EQ-5D-5L | Immediately post-intervention (up to 12 weeks)
  The EuroQol-5 Dimensions (EQ-5D-5L) is a measure of health-related quality of life. It consists of five items measuring five dimensions of health-related quality of life (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a vertical visual analogue scale measuring self-rated health.
EQ-5D-5L | 6 months post-intervention
  The EuroQol-5 Dimensions (EQ-5D-5L) is a measure of health-related quality of life. It consists of five items measuring five dimensions of health-related quality of life (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) and a vertical visual analogue scale measuring self-rated health.
PHQ-9 | Baseline
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item measure that rates the frequency of symptoms and is designed for screening, diagnosing, monitoring, and measuring the severity of depression.
PHQ-9 | Immediately post-intervention (up to 12 weeks)
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item measure that rates the frequency of symptoms and is designed for screening, diagnosing, monitoring, and measuring the severity of depression.
PHQ-9 | 6 months post-intervention
  The Patient Health Questionnaire-9 (PHQ-9) is a 9-item measure that rates the frequency of symptoms and is designed for screening, diagnosing, monitoring, and measuring the severity of depression.
Health Promoting Activities Scale | Baseline
  The HPAS is an 8-item measure of a person's estimation of the frequency with which they participate in a range of activities that promote or maintain health and well-being.
Health Promoting Activities Scale | Immediately post-intervention (up to 12 weeks)
  The HPAS is an 8-item measure of a person's estimation of the frequency with which they participate in a range of activities that promote or maintain health and well-being.
Health Promoting Activities Scale | 6 months post-intervention
  The HPAS is an 8-item measure of a person's estimation of the frequency with which they participate in a range of activities that promote or maintain health and well-being.
Patient Activation Measure (PAM) | Baseline
  The PAM is a 13-item measure that measures the spectrum of skills, knowledge, and confidence in patients and captures the extent to which people feel engaged and confident in managing their own health and care.
Patient Activation Measure (PAM) | Immediately post-intervention (up to 12 weeks)
  The PAM is a 13-item measure that measures the spectrum of skills, knowledge, and confidence in patients and captures the extent to which people feel engaged and confident in managing their own health and care.
Patient Activation Measure (PAM) | 6 months post-intervention
  The PAM is a 13-item measure that measures the spectrum of skills, knowledge, and confidence in patients and captures the extent to which people feel engaged and confident in managing their own health and care.
Parents' Assessment of Protective Factors | Baseline
  The PAPF is a 36-item measure that assesses protective factors identified in the development of the Strengthening Families evidence-based parenting programme. These protective factors are: parental resilience, social connections, concrete support in times of need, and support of children's social and emotional competence.
Parents' Assessment of Protective Factors | Immediately post-intervention (up to 12 weeks)
  The PAPF is a 36-item measure that assesses protective factors identified in the development of the Strengthening Families evidence-based parenting programme. These protective factors are: parental resilience, social connections, concrete support in times of need, and support of children's social and emotional competence.
Parents' Assessment of Protective Factors | 6 months post-intervention
  The PAPF is a 36-item measure that assesses protective factors identified in the development of the Strengthening Families evidence-based parenting programme. These protective factors are: parental resilience, social connections, concrete support in times of need, and support of children's social and emotional competence.
ICEpop CAPability measure for Adults (ICECAP-A) | Baseline
  The ICECAP-A is a 5-item measure of capability, which includes the following aspects of wellbeing found to be important to adults in the UK: attachment, stability, achievement, enjoyment, and autonomy. A set of UK utility values is available for the ICECAP-A, enabling it to be used in economic evaluations.
ICEpop CAPability measure for Adults (ICECAP-A) | Immediately post-intervention (up to 12 weeks)
  The ICECAP-A is a 5-item measure of capability, which includes the following aspects of wellbeing found to be important to adults in the UK: attachment, stability, achievement, enjoyment, and autonomy. A set of UK utility values is available for the ICECAP-A, enabling it to be used in economic evaluations.
ICEpop CAPability measure for Adults (ICECAP-A) | 6 months post-intervention
  The ICECAP-A is a 5-item measure of capability, which includes the following aspects of wellbeing found to be important to adults in the UK: attachment, stability, achievement, enjoyment, and autonomy. A set of UK utility values is available for the ICECAP-A, enabling it to be used in economic evaluations.
Service and Resource Use questionnaire | Baseline
  We will develop a resource use questionnaire in collaboration with parent carers. This will include health, social care, participant and broader societal resource use, and draw on measures in the Database of Instruments for Resource Use Management (DIRUM).
Service and Resource Use questionnaire | Immediately post-intervention (up to 12 weeks)
  We will develop a resource use questionnaire in collaboration with parent carers. This will include health, social care, participant and broader societal resource use, and draw on measures in the Database of Instruments for Resource Use Management (DIRUM).
Service and Resource Use questionnaire | 6 months post-intervention
  We will develop a resource use questionnaire in collaboration with parent carers. This will include health, social care, participant and broader societal resource use, and draw on measures in the Database of Instruments for Resource Use Management (DIRUM).
Programme Feedback Form | Immediately post-intervention (up to 12 weeks)
  We will collect feedback from treatment and control arm participants about the Healthy Parent Carer materials and delivery via a feedback form. All participants will be asked to complete the feedback form at 15 weeks post-randomisation.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Morris, DPhil, Principal Investigator — University of Exeter
Locations (6):
- United Kingdom (6):
  - Children's Hospice South West Little Harbour, St Austell, Cornwall
  - Learn Devon Bideford, Bideford, Devon
  - Orchard Manor School, Dawlish, Devon
  - Woodlands School, Plymouth, Devon
  - Torbay Parent Carer Forum, Torquay, Devon
  - The Beach Hotel, Minehead, Somerset

REFERENCES:
- [Background] Borek AJ, McDonald B, Fredlund M, Bjornstad G, Logan S, Morris C. Healthy Parent Carers programme: development and feasibility of a novel group-based health-promotion intervention. BMC Public Health. 2018 Feb 20;18(1):270. doi: 10.1186/s12889-018-5168-4. PMID 29458355
- [Background] Bjornstad G, Wilkinson K, Cuffe-Fuller B, Fitzpatrick K, Borek A, Ukoumunne OC, Hawton A, Tarrant M, Berry V, Lloyd J, McDonald A, Fredlund M, Rhodes S, Logan S, Morris C. Healthy Parent Carers peer-led group-based health promotion intervention for parent carers of disabled children: protocol for a feasibility study using a parallel group randomised controlled trial design. Pilot Feasibility Stud. 2019 Nov 23;5:137. doi: 10.1186/s40814-019-0517-3. eCollection 2019. PMID 31788323
- [Derived] Bjornstad G, Cuffe-Fuller B, Ukoumunne OC, Fredlund M, McDonald A, Wilkinson K, Lloyd J, Hawton A, Berry V, Tarrant M, Borek A, Fitzpatrick K, Gillett A, Rhodes S, Logan S, Morris C. Healthy Parent Carers: feasibility randomised controlled trial of a peer-led group-based health promotion intervention for parent carers of disabled children. Pilot Feasibility Stud. 2021 Jul 23;7:144. doi: 10.1186/s40814-021-00881-5. eCollection 2021. PMID 34301334
- See also: Healthy Parent Carers study website — http://sites.exeter.ac.uk/healthyparentcarers/